CLINICAL TRIAL: NCT06347302
Title: Study of Vitreoretinal Molecular Changes During Rhegmatogenous Retinal Detachment
Acronym: LIPIDRET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EID 2023
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Rhegmatogenous Retinal Detachments
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retinal detachment Group (Active Comparator)
  Interventions: Biological: Blood sampling; Other: vitreous sampling; Other: Sub-retinal fluid sampling; Other: Retinal tissue sampling
- Control group (Placebo Comparator)
  Interventions: Biological: Blood sampling; Other: vitreous sampling

INTERVENTIONS:
Biological: Blood sampling — Two tubes will be taken, the first tube (Tube 1) for specialised lipid analysis. The second tube (Tube 2) for routine biochemical analysis
Other: vitreous sampling — Intra-operative vitreous sampling: systematic collection of the vitreous humour during vitrectomy for vitreoretinal surgery such as retinal detachment, epiretinal membranes and macular holes.
Other: Sub-retinal fluid sampling — Sub-retinal fluid sampling consists of collecting the sub-retinal fluid that is systematically aspirated during retinal detachment surgery in order to dry the detached retina and allow retinopexy to be performed.
  Arms: Retinal detachment Group
Other: Retinal tissue sampling — cutting and aspiration of the retina using the vitreotome opposite the tear to allow access to the sub-retinal fluid.
  Arms: Retinal detachment Group

SUMMARY:
Retinal detachment is a condition with an estimated incidence of between 9.5 and 18.2 cases per 100,000 individuals.

It is an ophthalmological emergency that threatens visual acuity and requires surgery. However, despite satisfactory post-operative anatomical results, vitreoretinal proliferation and photoreceptor death can still have a negative impact on visual prognosis. These complications are still not fully understood.

A previous study carried out by the Eye, Nutrition and Cell Signalling team at the CSGA, comparing mouse models of retinal detachment with healthy control retinas, revealed an increase in pro-inflammatory cytokines and a change in retinal lipid abundance in detached retinas.

However, these results have yet to be confirmed in humans. Our main hypothesis is that the vitreous content of omega-3 PUFAs and proteins is altered during the onset of retinal detachment, since it reflects both intraocular inflammation and photoreceptor apoptosis.

We therefore wish to demonstrate that the protein and PUFA contents of the vitreous humour are different between eyes with retinal detachment and eyes not affected by retinal detachment after macular surgery (epiretinal membrane or macular hole). We would like to show that the vitreous PUFA content is lower in the macular surgery group due to the absence of photoreceptor apoptosis and the absence of dehiscence causing communication between the subretinal space (photoreceptors whose membranes are very rich in PUFAs) and the vitreous space. We also hope to identify changes in the protein composition of vitreous fluid in patients with retinal detachment, with overexpression of proteins involved in inflammation pathways.

In addition, we hypothesise that retinal omega-3 PUFA content is a factor influencing retino-vitreal proliferation and functional and anatomical recovery from retinal detachment. To this end, we will study the correlation between retinal PUFA-3 content and the clinical presentation and postoperative course of retinal detachment.

Finally, with the aim of identifying a serum marker for the prognostic evaluation of retinal detachment, we will use as a candidate a biomarker of retinal omega-3 PUFA content that we have developed in an Age-Related Macular Degeneration (AMD) model. We will analyse the correlation between this biomarker and levels of omega-3 PUFAs measured directly in the retina.

To do this, we will analyse intraoperative samples of vitreous humour, sub-retinal fluid and retinal fluid from patients undergoing vitrectomy for retinal detachment in the Ophthalmology Department of the Dijon University Hospital. A group of control patients will consist of patients operated on by vitrectomy for macular surgery (epiretinal membrane or macular hole) for whom a vitreous humour sample will also be taken.

Clinical information on the characteristics of the retinal detachment will be collected. During the consultation, the patient will be questioned about any history of dyslipidaemia and any current treatment, including the use of lipid-enriched food supplements. Post-operative follow-up with prospective collection of clinical and paraclinical data on anatomical and functional evolution will be carried out up to 6 months after the occurrence of retinal detachment.

A blood sample will be taken to establish a lipid profile in all patients. We will thus gain a better understanding of the changes in lipid and protein content in the vitreous humour, sub-retinal fluid and retina, and the demonstration of a link between the initial presentation and the postoperative anatomical and functional evolution of retinal detachment. This will provide a better understanding of the lipid-dependent mechanisms linked to inflammation and photoreceptor degeneration during retinal detachment, and will ultimately make it possible to develop new therapeutic strategies to improve visual prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject having given oral, free and informed consent to take part in the study
* Subjects with primary retinal detachment requiring vitrectomy (RD group) Or
* Subject requiring vitrectomy for macular surgery (primary epiretinal membrane or macular hole) (Control group)

Exclusion Criteria:

* Subject not affiliated to or not benefiting from national health insurance
* Pregnant, parturient or breast-feeding women
* Minors
* Subject to a measure of legal protection (curatorship, guardianship)
* Subjects of full age who are incapable or unable to express their consent
* Subject who has already participated in the study
* Subject with recurrent retinal detachment
* Subjects with an epiretinal membrane of secondary origin (OVCR, inflammation, diabetic retinopathy)
* Subject refusing blood sampling
* Subjects with pre-existing retinal pathology (vascular or degenerative retinopathy)
* People with diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Molecular content of fatty acids and proteins in the vitreous humour of eyes operated on for retinal detachment and eyes operated on for macular surgery | At the time of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France